CLINICAL TRIAL: NCT02914236
Title: A Prospective, Multi-Center Non-Randomized Study to Evaluate Treatment of Nasal Airway Obstruction Using the Aerin Medical Device
Brief Title: Treatment of Nasal Airway Obstruction Using the Aerin Medical Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP258
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2018-03-06 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Nasal Obstruction
Keywords: Nasal valve; Nasal airway obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vivaer Stylus (Experimental): Intervention: Procedure: thermal treatment of submucosal tissue including cartilage in the internal nasal valve area
  Interventions: Device: Vivaer Stylus

INTERVENTIONS:
Device: Vivaer Stylus — Delivery of low-power, temperature-controlled, radiofrequency energy to the tissues of the internal nasal valve area
  Other Names: Aerin Medical Device

SUMMARY:
Evaluation of the Aerin Medical Device used for the treatment of nasal obstruction.

DETAILED DESCRIPTION:
This is a non-significant risk, prospective, multi-center, non-randomized study to evaluate the safety and efficacy of the Aerin Medical device (Vivaer Stylus) when used to deliver radiofrequency (RF) energy to the nasal valve area to improve symptoms in those diagnosed with nasal airway obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for nasal obstruction and willing to undergo an office-based procedure
* Nasal Obstruction Symptom Evaluation (NOSE) score of ≥ 60 at Baseline
* Nasal valve is a primary or significant contributor to the subject's nasal obstruction as determined by the study investigator (based on clinical presentation, physical examination, nasal endoscopy, etc.) and the subject has a positive response to any of the following temporary measures (based on patient history or office exam):
* Use of external nasal dilator strips (e.g., Breathe Right Strips)
* Q-Tip test (manual intranasal lateralization)
* Use of nasal stents
* Cottle Maneuver (manual lateral retraction of the cheek)

Exclusion Criteria:

* Prior surgical treatment of the nasal valve
* Rhinoplasty, septoplasty, inferior turbinate reduction or other surgical nasal procedures within the past twelve (12) months
* Chronic sinusitis, recurrent sinusitis, or allergies leading to nasal obstruction
* Septal deviation, turbinate hypertrophy, polyps, or ptotic nose tip believed to be a significant contributor to the subject's nasal obstruction symptoms
* Known or suspected allergies or contraindications for any general or local anesthetic agents and / or any antibiotic medications
* Known or suspected to be pregnant, or is lactating
* Other medical conditions which in the opinion of the investigator could predispose the subject to poor wound healing or increased surgical risk

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wolf, MD, Study Director — Aerin Medical; Ofer Jacobowitz, MD, PhD, Principal Investigator — Mount Sinai Hospital, New York, NY
Locations (9):
- United States (9):
  - Central California Clinical Research, Fresno, California
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - ENT and Allergy Associates, LLP, Oradell, New Jersey
  - ENT and Allergy Associates, LLP, Bayside, New York
  - ENT and Allergy Associates, LLP, New Hyde Park, New York
  - ENT and Allergy Associates, LLP, New York, New York
  - ENT and Allergy Associates, LLP, Staten Island, New York
  - Piedmont Ear, Nose and Throat Associates, Winston-Salem, North Carolina
  - Ear, Nose and Throat Associates of Texas, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in the specialist's clinic with symptoms associated with nasal airway obstruction were approached for possible participation. Following completion of the informed consent process, baseline evaluation was conducted.
Pre-assignment Details: Four potential subjects failed to meet one or more of the inclusion/exclusion criteria. One additional subject met all criteria, but other health issues precluded commitment to the study.
Period: Overall Study
Arm/Group | Vivaer Stylus
Started (Underwent procedure) | 50
4-week Follow-up Visit | 50
12-week Follow-up Visit | 50
26-week Follow-up Visit | 49
Completed | 49
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vivaer Stylus
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 50
Nasal Obstruction Symptom Evaluation (NOSE) score [Mean (Standard Deviation); unit: units on a scale] — The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increased symptoms/symptom severity.
  units on a scale | 79.9 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in NOSE Score
Description: Mean change in Nasal Obstruction Symptom Evaluation (NOSE) score from baseline to 26 weeks post-study procedure. Improvement (baseline score - 26-week score) is signified by a positive value.
  The Nasal Obstruction Symptom Evaluation (NOSE) scale is a validated disease-specific health status outcomes instrument, used to assess severity of nasal obstruction symptoms. Score ranges from 0 to 100. Higher scores indicate increased symptoms/symptom severity.
Time Frame: Baseline, 26 weeks
Population: Does not include subject lost-to-follow-up prior to the 26-week follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vivaer Stylus
Number analyzed (Participants) | 49
units on a scale | 54.8 (21.9)
Statistical Analysis 1: Comparison: Vivaer Stylus; Test type: Superiority; p < 0.0001, t-test, 2 sided; Hypothesis was that the mean improvement in NOSE score exceeded 15 points

2. Secondary Outcome: NOSE Responder Rate
Description: Percent subjects who are responders to therapy; responder is defined as a treated subject who experiences at least a 15-point improvement in NOSE score from baseline to 26 weeks post treatment.
Time Frame: Baseline, 26 weeks
Population: Does not include subject lost-to-follow-up prior to 26-week follow-up
Measure: Number (95% Confidence Interval); unit: percentage of treated subjects
Arm/Group | Vivaer Stylus
Number analyzed (Participants) | 49
percentage of treated subjects | 93.9 [83.5 to 97.9]
Statistical Analysis 1: Comparison: Vivaer Stylus; Test type: Superiority; p < 0.0001, binomial test; Success threshold required at least 55% of subjects to be responders

3. Secondary Outcome: Percentage of Participants With Treatment-Related Adverse Events (Safety)
Description: Characterization of the type and frequency of treatment-related adverse events reported during or following the study procedure, throughout the follow-up period.
Time Frame: Baseline through 26 weeks
Population: All treated subjects
Measure: Number; unit: percentage of subjects having an event
Arm/Group | Vivaer Stylus
Number analyzed (Participants) | 50
percentage of subjects having an event | 20

4. Other Pre Specified Outcome: Subject-reported Pain Related to the Study Procedure, as Reported on 100mm Visual Analog Scale
Description: Procedure-related pain as reported by the subject using a 100mm Visual Analog Scale (VAS), immediately post-procedure and at the 4-week follow-up visit. Higher scores indicate more severe pain.
  The Pain VAS is presented to the subject as a 100mm line anchored on each end by verbal descriptors: 0 = no pain and 100 = worse pain imaginable. The distance between 0 and the vertical mark made by the subject is measured and the result is expressed in millimeters.
Time Frame: Immediately after study procedure, 4-weeks
Population: All treated subjects were asked to rate the pain level in each of their nostrils immediately following the treatment procedure and at the 4-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Nostrils
Arm/Group | Vivaer Stylus
Number analyzed (Participants) | 50
Number analyzed (Nostrils) | 99
units on a scale
  Post-Procedure, left nostril: number analyzed (Nostrils) | 50
  Post-Procedure, left nostril | 28.7 (26.0)
  Post-Procedure, right nostril: number analyzed (Participants) | 49
  Post-Procedure, right nostril: number analyzed (Nostrils) | 49
  Post-Procedure, right nostril | 26.9 (23.9)
  4-week visit, left nostril: number analyzed (Nostrils) | 50
  4-week visit, left nostril | 8.9 (16.0)
  4-week visit, right nostril: number analyzed (Nostrils) | 50
  4-week visit, right nostril | 8.7 (14.5)

5. Other Pre Specified Outcome: Subject Satisfaction
Description: Study-specific survey to assess patient satisfaction with the discomfort of the procedure and recovery period, as well as their perceived results. The survey included 5 questions related to tolerability of the procedure, ease of recovery, change in breathing, satisfaction with treatment, and willingness to recommend treatment. Each question was scored on a 10-point scale, with 1 indicating the most negative response to the question (e.g., "very bad", "much worse", or "very dissatisfied") and 10 indicating the most favorable rating (e.g., "hardly noticeable", "much better", or "very satisfied"). Each question was individually scored and reported.
Time Frame: 26 weeks
Population: Does not include subject lost-to-follow-up prior to 26-week follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vivaer Stylus
Number analyzed (Participants) | 49
units on a scale
  Q1 - Procedure tolerability | 7.3 (2.4)
  Q2 - Ease of recovery | 8.3 (1.7)
  Q3 - Breathing through nose | 8.3 (1.8)
  Q4 - Satisfaction with treatment | 8.4 (2.1)
  Q5 - Likely to recommend to others | 8.7 (2.1)

ADVERSE EVENTS:
Time Frame: From procedure through 26-week follow-up visit
Description: All subjects were queried for adverse events after the procedure and at each follow-up visit. Details of events were documented on a standardized case report form. Anticipated observations in the treatment area (such as swelling, redness, or crusting related to the treatment of tissue with radiofrequency energy) were not considered adverse events unless they required mitigation or were greater in severity, duration or degree of incidence than expected.
Arm/Group | Vivaer Stylus
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 18/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaer Stylus (N=50)
Appendicitis (Gastrointestinal disorders) | 1 (1) — unrelated to device or procedure
Balance disorder (Nervous system disorders) | 1 (1) — Recurrence of multiple sclerosis symptoms; unrelated to device or procedure
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaer Stylus (N=50)
nasopharyngitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Nasal edema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Presyncope (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of study results shall be made in conjunction with the results from all clinical study centers participating in the multicenter study. If results of the multi-center study have not been published in full within 18 months after completion of the study, investigator shall be free to publish results. Investigator agrees to submit all proposed publications to the sponsor at least 60 days prior submission; the company has the right to comment.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT02914236/Prot_SAP_000.pdf